CLINICAL TRIAL: NCT00484731
Title: Investigating the Effect of Intra-operative Infiltration With Local Anaesthesia on the Development of Chronic Postoperative Pain After Inguinal Hernia Repair. A Randomized Placebo Controlled Triple Blinded and Group Sequential Study Design
Brief Title: Effect of Intraoperative Infiltration With Bupivacain on the Development of Chronic Pain After Inguinal Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Luzerner Kantonsspital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 585; ISRCTN pending
Record Dates: First submitted 2007-06-07; First posted 2007-06-11 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Sodium Chloride; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Injection with Saline (Placebo Comparator): Injection with Saline instead of Bupivacain
  Interventions: Procedure: Infiltration with Saline
- Injection with Bupivacaine (Active Comparator): Injection with Bupivacaine
  Interventions: Procedure: Infiltration with Bupivacaine

INTERVENTIONS:
Procedure: Infiltration with Saline — Infiltration with Bupivacaine according to protocol
  Arms: Injection with Saline
Procedure: Infiltration with Bupivacaine
  Arms: Injection with Bupivacaine

SUMMARY:
The effect of intraoperative infiltration of the operation site with bupivacain on the development of chronic pain is the object of our trial. We hypothesize that the occurrence of chronic pain in the goup of patients receiving the infiltration will be 50% less than in the placebo group receiving normal saline. The study is a randomized controlled triple blinded trial with a sequential study design.

DETAILED DESCRIPTION:
264 patients scheduled for an inguinal hernia repair using one of three procedures (Lichtenstein, Barwell and TEP = total extraperitoneal hernioplasty) are being randomly allocated intra-operatively into two groups. Group I patients receive a local injection of 20ml Carbostesin® 0.25% at the end of the operation according to a standardised procedure. Group II patients get a 20 ml placebo (0.9% Saline) injection. We use pre-filled identically looking syringes for blinded injection, i.e. the patient, the surgeon and the examinator who performs the postoperative clinical follow-ups remain unaware of group allocation. The primary outcome of the study is the occurrence of developing chronic pain (defined as persistent pain at 3 months FU) measured by VAS and Pain Matcher® device (Cefar Medical AB, Lund, Sweden).

In addition to a sample size re-evaluation three interim analyses are planned after 120, 180 and 240 patients had finished their 3-months follow-up to allow for early study termination.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years) with primary or recurrent single or double sided symptomatic but not incarcerated inguinal hernias with an elective hernia repair are included.
* No other interventions (i.e. umbilical hernia) are allowed.
* Written informed consent needs to be obtained.

Exclusion Criteria:

* Patients with legal incompetence,
* Pregnant and nursing women,
* Patients with presence or history of active malignancy or systemic diseases,
* Under immunosuppressive treatment,
* With systemic or severe local inflammation or infection,
* With wound healing disorders and with physical or mental incapacity, which makes it impossible to obtain informed consent are excluded.
* As pacemakers interfere with the electrical stimulation of the Pain Matcher® and vice versa patients with pacemakers or other implanted electrical devices were also excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 404 (Actual)
Dates: Start 2006-07; Primary Completion 2011-12 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
occurrence of chronic pain | 3 months

SECONDARY OUTCOMES:
Level of Pain:Pain Matcher®,VAS;Areas of hyperalgesia,hypaesthesia Hospitalization:Length of stay (days) ASA-Classification Beginning of mobilisation (days) Return to work or normal activity (days and %) Quality of life (SF36) | one year

CONTACTS AND LOCATIONS:
Overall Officials: Jürg Metzger, Prof. Dr. med., Principal Investigator — Luzerner Kantonsspital
Locations (1):
- Kantonsspital Luzern, Lucerne, Switzerland

REFERENCES:
- [Derived] Honigmann P, Fischer H, Kurmann A, Audige L, Schupfer G, Metzger J. Investigating the effect of intra-operative infiltration with local anaesthesia on the development of chronic postoperative pain after inguinal hernia repair. A randomized placebo controlled triple blinded and group sequential study design [NCT00484731]. BMC Surg. 2007 Nov 6;7:22. doi: 10.1186/1471-2482-7-22. PMID 17986324